## FOREward Together: Training Peer Recovery Coaches to Promote Retention and Adherence to MOUD

NCT05098795

Approved Statistical Analysis Plan
Approved 7/31/2024

## **Data Analytic Plan**

Primary Outcomes: MOUD treatment retention and feasibility of intervention delivery.

Descriptive statistics will be used to characterize the sample. MOUD retention was defined *a priori* as return visits, measured for up to 24 weeks. We will calculate the percentage of participants still enrolled in the program over this period of time. Feasibility was defined, *a priori*, as the percent of patients who agreed to participate in the intervention. We will calculate the proportion of individuals who were screened eligible to the percent that engaged in the intervention, measured at study completion.

Secondary Outcomes: Intervention acceptability and intervention fidelity

Descriptive statistics will be examined for all secondary outcomes. Intervention acceptability was defined *a priori* as the percentage of patients enrolled who attend at least 75% of scheduled sessions. Intervention fidelity was defined *a priori* as the percentage of intervention elements delivered as intended. Following fidelity coding, we will calculate the number of accurately delivered components relative to the total number of coded components among a random selection of 20% of sessions.